CLINICAL TRIAL: NCT05566210
Title: Effects of Acupuncture on Ovarian Reserve Function and Pregnancy Outcomes in Women With Decreased Ovarian Reserve: a Multicenter Randomized Controlled Clinical Study
Brief Title: Effects of Acupuncture on Ovarian Function and Pregnancy Outcomes in Women With Decreased Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Cui Hong Zheng, Associate professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S266
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-09

CONDITIONS: Decreased Ovarian Reserve
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Active Comparator): Acupuncture was performed 2-3 times a week for 30 minutes each time for 3 months, starting from the 5th day of menstruation (spontaneous menstruation or drug withdrawal hemorrhaging menstruation)
  Interventions: Device: acupuncture
- Sham acupuncture group (Placebo Comparator): Sham acupuncture was performed 2-3 times a week for 30 minutes each time for 3 months, starting from the 5th day of menstruation (spontaneous menstruation or drug withdrawal hemorrhaging menstruation)
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: acupuncture — acupuncture
  Arms: Acupuncture group
Device: Sham acupuncture — Sham acupuncture
  Arms: Sham acupuncture group

SUMMARY:
The randomized, placebo-controlled multicenter trial is conducted in three centers in China. After screening and obtaining the signed informed consent, the participants are randomly divided into two groups: acupuncture group and sham acupuncture group.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women older than 18 years and younger than 40 years to undergo fresh IVF or self-pregnant;
2. AMH<1.1 ng/ml；
3. total AFC< 7；
4. 10 U/L<FSH< 25IU/L,或FSH/LH>2.6；
5. had a history of low ovarian response once, and the number of eggs obtained in IVF was less than 3 （at least two of the 2）3）4）5 ）items are required）；
6. Willing to accept randomized grouping, treatment arrangement and follow-up, and signing informed consent.

Exclusion Criteria:

Patients who met any of the following conditions were not included:

1. Severe abnormality of uterine cavity caused by adenomyosis, uterine fibroids, endometrial polyps, tuberculosis of the reproductive system, endometritis, abnormal endometrial thickness (HCG day of the previous IVF cycle is less than 7mm or greater than 14mm);
2. Patients with other endocrine diseases, such as thyroid disease, hyperprolactinemia, insulin resistance, diabetes, adrenal disease, etc., and poor control of hormone levels in the last 3 months;
3. Clearly diagnosed autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome, etc.;
4. Untreated hydrosalpinx;
5. Body mass index (BMI) higher than 28 kg/m;
6. The male or female chromosome abnormality;
7. People with previous history of acupuncture sickness;
8. Those who have previously participated in the study or are currently receiving acupuncture treatment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
AFC | on the 3rd day of menstruation
  Antral follicle count

SECONDARY OUTCOMES:
Blood levels of FSH, LH, E2 and AMH on the 3rd day of menstruation | on the 3rd day of menstruation
β-HCG positive pregnancy rate | Two weeks after ET or when menstruation expired for natural pregnancy
Clinical pregnancy rate | 4 weeks after ET or natural pregnancy: B ultrasonography was used to observe whether there were pregnant sac and cardiac tube pulsation in uterine cavity
Live birth rate | Gestation greater than 24 weeks and birth as a live fetus

CONTACTS AND LOCATIONS:
Overall Officials: Cuihong Zheng, Professor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital,Tongji medical college,HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No